CLINICAL TRIAL: NCT00182845
Title: Preventing Post-Operative Cognitive Decline
Brief Title: Donepezil in the Prevention of Post-Operative Cognitive Decline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IA0078
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Postoperative Complications; Delirium
Keywords: dementia; MCI; Aricept; Adverse Effects; Hospital Acquired Complications; Cognitive Impairment; Aging
MeSH Terms: conditions — Postoperative Complications; Delirium; Dementia; Cognitive Dysfunction | interventions — Donepezil

INTERVENTIONS:
Drug: Donepezil

SUMMARY:
The purpose of this study is to evaluate the feasibility of using Donepezil to prevent post-operative cognitive decline (POCD) among individuals aged 65 and older who have a baseline mild cognitive impairment (MCI) and are undergoing elective hip or knee replacement.

DETAILED DESCRIPTION:
Up to 65% of elderly patients undergoing hip or knee surgery suffer from declining brain function known as post-operative cognitive decline (POCD). These individuals often stay in the hospital longer, have more complications, and are more likely to die. Recent clinical studies have shown the potential benefit of enhancing the cholinergic system among patients with both Alzheimer's disease and / or vascular dementia. Donepezil is currently being used to treat memory loss in patients with Alzheimer's disease.

This study will recruit 30 cognitively impaired adults aged 65 or older who are scheduled to have elective hip or knee replacement surgery at University Hospital. Participants will be randomized to receive either a three to six week supply of Donepezil or a matching placebo approximately 4 weeks prior to surgery. This study will evaluate the effect of Donepezil on delirium incidence and severity during hospitalization, global cognitive function, length of hospitalization, site of discharge, and adverse drug effects.

All material to be collected will be from interviews, questionnaires, and medical chart review. Some will be at baseline, during hospitalization, and 12 weeks post hospitalization and others will be daily during hospitalization. The International Study of Post-Operative Cognitive Decline battery of tests will be used in assessment, as will the CogHealth computerized battery.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling individuals aged 65 or older
* Scheduled for elective hip or knee replacement at University Hospital
* Mild cognitive impairment, defined as:

  * MMSE total score of 27 or less;
  * normal performance of the activities of daily living tasks of the Bristol scale after excluding mobility related difficulties;
  * no chart-based dementia diagnosis; and
  * no history of ever being on dementia medications such as Memantine or any cholinesterase inhibitors
* Consent to participate in the study

Exclusion Criteria:

* Chart-based dementia diagnosis
* MMSE score greater than 27
* Difficulty performing the activities of daily living not related to mobility as measured by the Bristol scale
* Current or past history of receiving dementia medications such as Memantine or any cholinesterase inhibitors (Tacrine, Donepezil, Rivastigmine, or Galantamine)
* Metastatic cancer or other comorbid illnesses likely to reduce life expectancy to under 6 months
* Multiple trauma or pathological fractures requiring acute hip or knee replacement
* Aphasic, blind, or deaf
* Use of neuroleptics one month prior to surgery
* Allergy to donepezil
* Inability to read and complete study tests and forms
* Alcohol or drug dependence, defined as intake of more than 5 units of alcohol daily during the past 3 months
* Not expected to be discharged from hospital or able to complete the 3-month postoperative test
* Not competent to make medical decisions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30
Dates: Start 2005-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Changes in the International Study of Post-Operative Cognitive Decline (ISPOCD) and the CogHealth computerized battery tests at 1 week and 12 weeks after surgery

SECONDARY OUTCOMES:
Delirium status measured by the Confusion Assessment Method (CAM) and the Memorial Delirium Assessment Scale (MDAS) daily during the post-operative period
Global cognitive status assessed using the Mini Mental Status Exam (MMSE)
Length of stay in the hospital post-operatively
Discharge site
Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Malaz Boustani, MD, MPH, Principal Investigator — Regenstrief Institute, Indiana University Center for Aging Research
Locations (1):
- University Hospital, Clarian Health Partners, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Dodds C, Allison J. Postoperative cognitive deficit in the elderly surgical patient. Br J Anaesth. 1998 Sep;81(3):449-62. doi: 10.1093/bja/81.3.449. No abstract available. PMID 9861139
- [Background] Rasmussen LS. Defining postoperative cognitive dysfunction. Eur J Anaesthesiol. 1998 Nov;15(6):761-4. doi: 10.1097/00003643-199811000-00026. No abstract available. PMID 9884870
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Abildstrom H, Rasmussen LS, Rentowl P, Hanning CD, Rasmussen H, Kristensen PA, Moller JT. Cognitive dysfunction 1-2 years after non-cardiac surgery in the elderly. ISPOCD group. International Study of Post-Operative Cognitive Dysfunction. Acta Anaesthesiol Scand. 2000 Nov;44(10):1246-51. doi: 10.1034/j.1399-6576.2000.441010.x. PMID 11065205
- [Background] Johnson T, Monk T, Rasmussen LS, Abildstrom H, Houx P, Korttila K, Kuipers HM, Hanning CD, Siersma VD, Kristensen D, Canet J, Ibanaz MT, Moller JT; ISPOCD2 Investigators. Postoperative cognitive dysfunction in middle-aged patients. Anesthesiology. 2002 Jun;96(6):1351-7. doi: 10.1097/00000542-200206000-00014. PMID 12170047